CLINICAL TRIAL: NCT06908148
Title: SALACIA: Randomised Control Trial of SALvesAn Neutral Electrolysed Water Versus Conventional Management of Non-healing dIAbetic Foot Wounds
Brief Title: SALACIA: SALvesAn vs Conventional Management of dIAbetic Foot Wounds
Acronym: SALACIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L22044C
Record Dates: First submitted 2025-01-21; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-01

CONDITIONS: Foot Ulcers, Diabetic; Foot Ulcer Unhealed
Keywords: Foot Ulcers; Diabetic; Wound Healing; Electrolysed Water
MeSH Terms: conditions — Foot Ulcer

STUDY DESIGN:
Intervention Model Description: Randomised control trial to compare electrolysed water against conventional management of non-healing diabetic foot wounds
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electrolysed water (Experimental): Electrolysed water is a novel antiseptic produced by passing an electric current through a mixture of tap water and salt. Microbiocidal activity is due to the presence of hypochlorous acid at neutral Ph. Irrigation of chronic wounds reduces bacterial load and appears to encourage wound healing. We propose to compare electrolysed water against conventional management.
  Interventions: Device: Electrolysed water
- Conventional irrigant (Active Comparator): The irrigant (Prontosan™) that is currently 'in-use' in the conventional management of diabetic foot wounds
  Interventions: Device: Conventional irrigant

INTERVENTIONS:
Device: Electrolysed water — Electrolysed water is a novel antiseptic produced by passing an electric current through a mixture of tap water and salt. Microbiocidal activity is due to the presence of hypochlorous acid at neutral Ph. Irrigation of chronic wounds reduces bacterial load and appears to encourage wound healing. We propose to compare electrolysed water against conventional management.
  Arms: Electrolysed water
Device: Conventional irrigant — The irrigant (Prontosan™) that is currently 'in-use' in the conventional management of diabetic foot wounds
  Arms: Conventional irrigant

SUMMARY:
Increasing prevalence of diabetes mellitus has led to increasing numbers of chronic non-healing foot ulcers (wounds).

Electrolysed water is a novel antiseptic which reduces bacterial load and appears to encourage wound healing. The investigators propose to compare electrolysed water against conventional management.

DETAILED DESCRIPTION:
Increasing prevalence of diabetes mellitus has led to increasing numbers of chronic non-healing foot ulcers (wounds). These wounds are colonised with pathogens, including multi-drug resistant organisms. Despite repeated courses of antibiotics, subsequent management is difficult due to devascularisation of surrounding tissues and healing failures. Ultimately, patients may require amputation.

Electrolysed water is a novel antiseptic produced by passing an electric current through a mixture of tap water and salt. Microbiocidal activity is due to the presence of hypochlorous acid at neutral Ph. Irrigation of chronic wounds reduces bacterial load and appears to encourage wound healing. The investigators propose to compare electrolysed water against conventional management.

Patients who attend NHS podiatry clinics, and who enrol in the trial, will receive treatment of their wounds as-per routine care; the only difference is the irrigant used. Patients will be randomised to use either the in-use product (Prontosan™) or electrolysed water (Salvesan).

The inclusion criteria are:

* Adult diabetic patients (18-89 years)
* Chronic wounds (present for >=3 weeks since commencing Podiatry care)
* Non-healing (wounds that, in the view of the patient's Podiatrist, are not responding to standard treatment)
* Wounds that are >=5mm when measured in any direction The treatment phase will last for 12 weeks (or less, if complete healing achieved). All patients will be followed up at 20 weeks to assess recurrence. Primary composite end-point defined as time to complete healing or proportion achieving >50% healing if complete healing is not achieved.

Primary objective is to compare rapidity of wound healing. Secondary endpoints are surgical intervention, debridement, amputation, patient death.

Improved healing could potentially benefit patients who might otherwise progress to amputation. The investigators will monitor antimicrobial consumption in study patients throughout the trial. A final objective is to carry out an economic evaluation of electrolysed water vs Prontosan in the routine management of non-healing foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Adult diabetic patients (18-89 years)
* Chronic wounds (present for >=3 weeks since commencing Podiatry care)
* Non-healing (wounds that, in the view of the patient's Podiatrist, are not responding to standard treatment)
* Wounds that are >=5mm when measured in any direction

Exclusion Criteria:

* Patients lacking capacity to provide informed consent
* Patients with underlying terminal disease
* Patients with severe comorbidities, e.g. morbidly obese; uncontrolled diabetes (HbA1c > 97 mmol/mol); gangrene; chronic leg oedema/venous disease; end-stage renal disease; untreatable ischaemic heart disease; HIV; etc.
* Women who are pregnant or breastfeeding will be excluded from this trial.
* Women of child-bearing potential who are not using an acceptable form of contraception will be excluded from this trial.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of diabetic foot ulcers (wounds) that heal when irrigated using electrolysed water versus the proportion that heal when using the standard-of-care irrigant | From enrollment to 20 weeks
  This investigation seeks to determine whether irrigation of non-healing diabetic foot ulcers (wounds) using neutral electrolysed water (Salvesan) results in equivalent, or better, wound healing than the standard-of-care wound management irrigant (Prontosan® Solution).
  The primary outcome measure is the condition of the wound at the end of the study, with composite end-points defined as:
  (A) - for wounds that heal completely within the 12-week follow up period, the associated time to completely heal
  (B) - for wounds that do not completely heal, the number with >50% healing of initial lesion at 12 weeks (defined as surface area in mm2 as measured using the standard methodology used within the Diabetic Podiatry service).
  The proportions of wounds that heal [(A)- completely / (B) - with >50% healing] using each irrigant will be compared statistically to assess whether there is any difference in the proportion healed using electrolysed water versus standard-of-care irrigant.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lewis, Study Director — Aqualution